CLINICAL TRIAL: NCT03458546
Title: Phase Ib Clinical Trial of Roflumilast Added to Standard Chemoimmunotherapy for High-risk Diffuse Large B-cell Lymphoma
Brief Title: Study of Roflumilast in Combination With Standard Chemotherapy for High-risk Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 17-0087; 18-073H (Other: UTHSA IRB)
Record Dates: First submitted 2018-02-19; First posted 2018-03-08 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-02

CONDITIONS: Lymphoma, B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Roflumilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Roflumilast and R-CHOP (Experimental)
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — All patients will receive R-CHOP therapy at standard doses according to the standard preparation and infusion procedures of each investigational site, which is to be repeated every 21 days for a total of 6 cycles. All patients will receive a fixed oral dose of one 500 microgram (μg) tablet per day with or without food for all 21 days of each cycle, which will amount to a total of 126 doses of roflumilast.
  Other Names: Daliresp

SUMMARY:
This study is a phase Ib, single arm, open label clinical trial that will enroll patients with untreated diffuse large B-cell lymphoma (DLCBL) at moderate or high risk for poor outcome

DETAILED DESCRIPTION:
This study is a phase Ib, single arm, open label clinical trial that will enroll patients with untreated diffuse large B-cell lymphoma (DLCBL) at moderate or high risk for poor outcome, defined as an NCCN-IPI score of 2 or higher. Each patient's disease will be biologically characterized at baseline. Enrolled patients will receive chemoimmunotherapy with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP), administered every 21 days for 6 cycles, which is the standard of care. In addition, all patients will receive the study drug, roflumilast, at the standard dose of 500 μg by mouth once daily, throughout the 18-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older.
* Pathologically proven diffuse large B-cell lymphoma.
* No prior systemic therapy for lymphoma.
* NCCN-IPI risk score of 2 or higher.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy of ≥3 months.
* Ann Arbor stage II-IV
* Measurable disease, meaning at least 1 lymph node or other lymphomatous lesion with a long axis of ≥1.5 cm by CT imaging, and at least one FDG-avid lesion by FDG-PET scan.
* Left ventricular ejection fraction of at least 45% by either echocardiography or radionucleotide angiography.
* Ability to swallow oral tablets without difficulty.
* All subjects with preserved reproductive potential must agree to practice abstinence or employ contraceptive measures for the duration of treatment and for 4 weeks following final dosing. All male subjects are considered to have reproductive potential. Female subjects of reproductive potential are those who: 1) are not at least 50 years old and have no menses for 24 consecutive months; or 2) have not been rendered surgically sterile (having undergone hysterectomy and/or bilateral salpingo-oophorectomy). Female subjects of reproductive potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin ([hCG]) within 7 days of first day of drug dosing.
* Meet the following clinical laboratory requirements: - Creatinine clearance ≥30 ml/min by Cockcroft-Gault formula ; - Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (unless indirect bilirubin is elevated due to Gilbert's syndrome or hemolysis); - AST and ALT≤ 3 × ULN; - Platelet count ≥ 50,000/μL, with or without transfusion support; - ANC ≥ 1000/μL, with or without chronic granulocyte growth factor support; - Hemoglobin ≥8 g/dL, with or without transfusion support.

Exclusion Criteria:

* Allergy or intolerance to roflumilast.
* Any active malignancy other than DLBCL
* Prior allogeneic bone marrow transplant within 12 months of screening date.
* Prior autologous stem cell transplant within 6 months of screening date.
* Immunotherapy, chemotherapy, radiotherapy, or investigational therapy within 6 months prior to drug dosing.
* Active central nervous system (CNS) involvement by lymphoma, including untreated symptomatic epidural disease
* Active uncontrolled infection.
* Clinically documented history of severe depression and/or suicidal thoughts or behavior.
* Uncontrolled illness including but not limited to: symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV heart failure), unstable angina pectoris, uncontrolled cardiac arrhythmia, and psychiatric illness that would limit compliance with study requirements.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty and/or stent placement within 6 months prior to study drug dosing.
* History of another active cancer within 2 years prior to study drug dosing, excluding adequately treated basal cell or squamous cell carcinoma of the skin, cervical cancer in situ, or other adequately treated in situ carcinoma.
* History of major surgery within 3 weeks or minor surgery within 1 week of roflumilast administration. Major surgery includes, for example, any open or laparoscopic entry into a body cavity, or operative repair of fracture; minor surgery includes, for example, open surgical biopsy of palpable/superficial lymph node, or placement of vascular access device.
* Other medical or psychiatric illness or organ dysfunction, which in the opinion of the investigator, would either compromise the subject's safety or interfere with the evaluation of the safety of the study agent.
* Corrected QT interval (QTc) prolongation (defined as a QTc >450 ms for males and >470 ms for females [Fridericia's correction]) or other clinically significant ECG abnormalities as assessed by the investigator.
* Patients known to be HIV-positive must not have multi-drug resistant HIV infection, CD4 counts < 150/μl or other concurrent AIDS-defining conditions. Serologic screening for HIV is required within the 6 months prior to study enrollment.
* Patients positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C-virus ribonucleic acid (HCV RNA), unless both AST and ALT≤1.25 x ULN and there is no known history of chronic active hepatitis. Serologic screening for hepatitis B and C testing is required within the 6 months prior to study enrollment.
* Patients with moderate or severe liver impairment, as defined by a Child-Pugh class of B or C.
* Women who are pregnant or breastfeeding.
* Current use of any of the following medications: boceprevir, carbamazepine, ciprofloxacin, cobicistat, conivaptan, enzalutamide, fluvoxamine, itraconazole, ketoconazole, mitotane, phenytoin, posaconazole, rifampin, ritonavir, St. John's Wort, telaprevir, voriconazole, or zafirlukast.
* Current use of non-nucleoside reverse transcriptase inhibitors (NNRTI) including efavirenz, rilpivirine, etravirine, delavirdine, nevirapine, and lersivirine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
To evaluate adverse drug reactions and toxicities as evaluated by NCI CTCAE using the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03 | Measured every 3 weeks for 21 day cycles for the duration of study treatment, estimated to be less than one year

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo E Diaz Duque, MD, Principal Investigator — Mays Cancer Center, UT Health San Antonio; Ricardo Aguiar, MD, PhD, Principal Investigator — Mays Cancer Center, UT Health San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duque AED, Ferrari PSSM, Ethiraj P, Jaafar C, Qiu Z, Holder K, Butler MJ, Huelgas-Morales G, Karnad A, Dahia PLM, Aguiar RCT. First-Line Combination of R-CHOP with the PDE4 Inhibitor Roflumilast for High-Risk DLBCL. Cancers (Basel). 2024 Nov 18;16(22):3857. doi: 10.3390/cancers16223857. PMID 39594812